CLINICAL TRIAL: NCT00006234
Title: A Phase I/II Study of 166Ho-DOTMP With Peripheral Blood Progenitor Cell Support for Refractory or Recurrent Ewing's Sarcoma Family of Tumors With Bone Disease
Brief Title: Holmium Ho 166 DOTMP Followed by Peripheral Stem Cell Transplantation in Treating Patients With Metastatic Ewing's Sarcoma or Rhabdomyosarcoma That Has Spread to the Bone
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1474.00; FHCRC-1474.00; CHMC-S-6007; NCI-G00-1842; CDR0000068159 (Registry Identifier: PDQ)
Record Dates: First submitted 2000-09-11; First posted 2003-01-27 (Estimated); Last update posted 2011-12-01 (Estimated); Status verified 2011-11

CONDITIONS: Metastatic Cancer; Sarcoma
Keywords: recurrent childhood rhabdomyosarcoma; recurrent adult soft tissue sarcoma; adult rhabdomyosarcoma; bone metastases; previously treated childhood rhabdomyosarcoma; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; stage IV adult soft tissue sarcoma
MeSH Terms: conditions — Neoplasm Metastasis; Sarcoma; Rhabdomyosarcoma; Neuroectodermal Tumors, Primitive, Peripheral | interventions — Peripheral Blood Stem Cell Transplantation; holmium-1,4,7,10-tetraazacyclododecane-N,N',N'',N'''-tetrakis(methylenephosphonic acid)

INTERVENTIONS:
Procedure: peripheral blood stem cell transplantation
Radiation: holmium Ho 166 DOTMP

SUMMARY:
RATIONALE: Radioactive drugs, such as holmium Ho 166 DOTMP, may carry radiation directly to cancer cells and not harm normal cells. Peripheral stem cell transplantation may be able to replace stem cells that were destroyed by the radioactive drug.

PURPOSE: This Phase I/II trial is studying the effectiveness of holmium Ho 166 DOTMP followed by peripheral stem cell transplantation in treating patients who have metastatic Ewing's sarcoma or rhabdomyosarcoma that has spread to the bone.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dosimetry of holmium Ho 166 DOTMP in patients with metastatic Ewing's sarcoma family of tumors or rhabdomyosarcoma with bone metastases.
* Provide treatment with holmium Ho 166 DOTMP for these patients.
* Determine the toxicity and pharmacokinetics of this drug in these patients.
* Determine the change in tumor cell content in peripheral blood and bone marrow after treatment with this drug in these patients.

OUTLINE: Patients receive a trace dose of holmium Ho 166 DOTMP IV over 10 minutes on day -7 and an assigned dose over 10 minutes on day 0. Autologous peripheral blood stem cells are infused on days 7-10.

Patients are followed at least weekly for 4 weeks and then monthly for 1 year or until disease progression.

PROJECTED ACCRUAL: A total of 4 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed Ewing's sarcoma family of tumors or rhabdomyosarcoma with bone metastases

  * Refractory to conventional therapy OR
  * Responsive to conventional therapy with osseous metastases at diagnosis that are extensive enough to preclude concurrent radiotherapy to all sites
* Soft tissue, pulmonary, and/or bone marrow metastases in addition to cortical bone allowed

  * Extraosseous sites of disease allowed if amenable to surgical resection or external beam radiotherapy
* No patients under 10 years old with embryonal rhabdomyosarcoma
* Adequate peripheral blood stem cells stored

  * At least 2,500,000 CD34+ cells/kg
* No impending bone fracture or spinal cord compression

PATIENT CHARACTERISTICS:

Age:

* 12 and over

Performance status:

* 0-2

Life expectancy:

* At least 2 months

Hematopoietic:

* Absolute neutrophil count at least 1,000/mm^3
* Platelet count at least 75,000/mm^3 (transfusion independent)
* Hemoglobin at least 10.0 g/dL (RBC transfusion allowed)

Hepatic:

* Bilirubin no greater than 1.5 times normal
* SGOT no greater than 2.5 times normal

Renal:

* Radioisotope glomerular filtration rate, iothalamate clearance, or creatinine clearance at least 60 mL/min

Other:

* No uncontrolled infection
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Recovered from prior immunotherapy
* At least 3 months since prior bone marrow or peripheral blood stem cell transplantation (6 months for total body irradiation conditioning) and recovered
* At least 1 week since prior cytokines
* No immunomodulators during and for at least 4 weeks after study
* No concurrent cytokines

Chemotherapy:

* At least 3 weeks since prior chemotherapy (6 weeks for nitrosoureas) and recovered
* No more than 3 prior systemic chemotherapy regimens
* No systemic chemotherapy during and for at least 4 weeks after study

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* See Biologic therapy
* Recovered from prior radiotherapy
* No prior maximum tolerable radiotherapy (greater than 30 Gy) to the spinal cord
* No prior therapeutic doses of bone-seeking radiopharmaceutical (e.g., samarium Sa 153 lexidronam pentasodium EDTMP)
* No radiotherapy during and for at least 4 weeks after study

  * Local radiotherapy to any tumor site allowed provided at least 1 evaluable lesion is untreated

Surgery:

* See Disease Characteristics
* No surgical resection of all bone metastases evaluable by PET during and for 1 month after study

Other:

* At least 4 weeks since prior bisphosphonates

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-11; Study Completion 2006-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Hawkins, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States